CLINICAL TRIAL: NCT01601132
Title: An Open-Label, One Sequence, Pharmacokinetic Drug Interaction Study of Colchicine and Theophylline in Healthy Subjects
Brief Title: Drug Interaction Study of Colchicine and Theophylline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-11-4001; U1111-1141-7355 (Registry Identifier: WHO)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: pharmacokinetics; colchicine; theophylline
MeSH Terms: interventions — Theophylline; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- theophylline (Experimental): 300mg (80mg/15ml elixir) theophylline
  Interventions: Drug: theophylline
- Colchicine (Experimental): colchicine 0.6mg by mouth twice daily on Days 5-19, co-administered with theophylline 300mg (80mg/15ml) on the morning of Day 19
  Interventions: Drug: colchicine

INTERVENTIONS:
Drug: theophylline — 300mg (80mg/15ml elixir)
  Other Names: Elixophyllin®
  Arms: theophylline
Drug: colchicine — colchicine 0.6mg by mouth twice daily on Days 5-19, co-administered with theophylline 300mg (80mg/15ml) on the morning of Day 19
  Other Names: COLCRYS®
  Arms: Colchicine

SUMMARY:
Colchicine is a supressor of hepatic CYP1A2 and theophylline is a sensitive CYP1A2 probe substrate. When the two are co-administered the potential exists for a clinically significant drug interaction. This study aims to determine the effect of steady-state colchicine on the pharmacokinetics of theophylline administered as a single dose. A secondary goal is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the entire study period.

DETAILED DESCRIPTION:
Colchicine is a supressor of hepatic CYP1A2 and theophylline is a sensitive CYP1A2 probe substrate. When the two are co-administered the potential exists for a clinically significant drug interaction. This study aims to determine the effect of steady-state colchicine on the pharmacokinetics of theophylline administered as a single dose. After a fast of at least 10 hours, thirty healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one dose of 300mg (80mg/15ml concentrate) theophylline (theophylline elixir) on Day 1. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately determine the pharmacokinetics of theophylline. Blood sampling will then continue on a non-confined basis on days 2-3. A four day washout period will be completed after the theophylline dose on Day 1 and prior to administration of the first colchicine dose on Day 5. Participants will return to the clinic on days 5-18 for non-confined dosing of colchicine (1x0.6mg twice daily every 12 hours). Administered dosing on these days will not necessarily be in a fasted state. Co-administration of a single 300mg dose of theophylline (80mg/15ml) and colchicine (1x0.6mg) will occur on the morning of Day 19 following a fast of at least 10 hours. Twelve hours later, subjects will receive the last dose of colchicine (1x0.6mg). Blood samples will be drawn from all participants before dosing on Day 19 and for 24 hours post-dose on a confined basis at times sufficient to adequately determine the pharmacokinetics of theophylline. Blood sampling will then continue on a non-confined basis on days 20 and 21. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to dosing and at approximately 1, 2, and 3 hours following drug administration on Days 1, 5 (after the morning dose) and 19. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non smoking and non-pregnant (postmenopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive; hemoglobin greater than or equal to 11.5g/dL

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or donation of plasma
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* Subjects who test positive for drugs of abuse or alcohol at screening or check-in
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease or active sexually transmitted disease
* History of neuropathy or muscle disorders, peptic ulcer disease, clinically significant cardiac arrhythmias, seizure disorder, and low white blood cell count or other bone marrow disorders
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* History of allergy or sensitivity to colchicine or theophylline or aminophylline
* Subjects who have had a tattoo or body piercing within 30 days prior to administration of study drug
* Subjects with irritable bowel syndrome, chronic diarrhea or other chronic gastro-intestinal problems
* Subjects who are lactose intolerant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, M.D., Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- Worlwide Clinical Trials Drug Development Solutions, Clinical Research Services, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the USA from 11 June 2012 to 01 July 2012.
Pre-assignment Details: Thirty non-smoking, adult male and female volunteers (ages 18 to 45 years) were enrolled in this single group study.
Groups:
- Theophylline + Colchicine: Theophylline 300 mg, solution, orally, on Day 1, then colchicine 0.6 mg tablets, orally, twice daily on Days 5-18, then theophylline 300 mg, solution, orally together with colchicine 0.6 mg, tablet, orally on Day 19 followed by a last dose of colchicine 0.6 mg, tablet, orally, 12 hours later.
Period: Overall Study
Arm/Group | Theophylline + Colchicine
Started | 30
Completed | 28
Not Completed | 2
Not completed — Patient withdrew consent | 1
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Theophylline + Colchicine
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 4
  White | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 7
Region of Enrollment [Number; unit: Participants]
  United States | 30
Tobacco history [Number; unit: Participants]
  Never used tobacco | 26
  Past smoker or has used other forms of tobacco | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Theophylline
Description: The time to each the maximum or peak concentration of theophylline in the plasma, after a single dose on Day 1, and after a single dose on Day 19, following 14 days of colchicine dosing.
Time Frame: Day 1 and Day 19 blood samples drawn pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours after dose administration.
Population: The pharmacokinetic (PK) population is defined as any participant who took a single dose of study medication and had sufficient blood sampling to characterize the non-compartmental PK parameters. Patients with available data are included in the analysis.
Measure: Median (Full Range); unit: hours
Groups:
- Theophylline: Theophylline 300 mg, solution, orally, on Day 1.
- Theophylline + Colchicine: Theophylline 300 mg, solution, orally together with colchicine 0.6 mg, tablet, orally on Day 19 followed by a last dose of colchicine 0.6 mg, tablet, orally, 12 hours later.
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
hours | 1.25 [0.25 to 4.00] | 1.5 [0.25 to 4.00]
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Test type: Superiority or Other; p = 0.5663, Wilcoxon (Mann-Whitney) — Significant difference defined a priori as p < 0.05

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Theophylline
Description: The maximum or peak concentration of theophylline in the plasma, after a single dose on Day 1, and after another single dose on Day 19 following 14 days of colchicine dosing.
Time Frame: as for outcome 1
Population: The pharmacokinetic (PK) population is defined as any participant who took a single dose of study medication and had sufficient blood sampling to characterize the non-compartmental PK parameters.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
μg/mL | 11.0 (2.16) | 11.7 (2.79)
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Analysis of variance (ANOVA) was performed on the log-transformed Cmax to calculate least squares mean (LSM) for each treatment. The ANOVA model included sequence, treatment, and treatment within a sequence as fixed effects, and participant as a random effect. The criterion for demonstrating a lack of a clinically significant interaction is a 90% CI for the ratio for AUC0-t, (AUC0-∞), and Cmax to be within the 0.80 to 1.25 interval, representing a maximum of 20% difference between treatments; Test type: Superiority or Other; ANOVA; Ratio (%) (Test/Reference) = 105.86, 90% CI 2-sided [101.77 to 110.12] — Ratio (theophylline+colchicine/theophylline) of LSMs calculated using the exponentiation of the difference between treatment LSM from the log-transformed Cmax, expressed as a percentage relative to the reference treatment

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time of the Last Quantifiable Concentration[AUC(0-t)]
Description: The area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule for theophylline.
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: hours*μg/mL
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
hours*μg/mL | 155.6 (34.86) | 164.0 (40.01)
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Analysis of variance (ANOVA) was performed on the log-transformed AUC(0-t) to calculate least squares mean (LSM) for each treatment. The ANOVA model included sequence, treatment, and treatment within a sequence as fixed effects, and participant as a random effect. The criterion for demonstrating a lack of a clinically significant interaction is a 90% CI for the ratio for AUC0-t, AUC0-∞, and Cmax to be within the 0.80 to 1.25 interval, representing a maximum of 20% difference between treatments; Test type: Superiority or Other; ANOVA; Ratio (%) (Test/Reference) = 105.63, 90% CI 2-sided [101.81 to 109.59] — Ratio (theophylline+colchicine/theophylline) of LSMs calculated using the exponentiation of the difference between treatment LSM from the log-transformed AUC(0-t)], expressed as a percentage relative to the reference treatment

4. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. [AUC(0-∞)] was calculated as the sum of AUC (0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant for theophylline.
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: hours*μg/mL
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
hours*μg/mL | 180.7 (62.30) | 185.7 (54.46)
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Analysis of variance (ANOVA) was performed on the log-transformed AUC(0-∞) to calculate least squares mean (LSM) for each treatment. The ANOVA model included sequence, treatment, and treatment within a sequence as fixed effects, and participant as a random effect. The criterion for demonstrating a lack of a clinically significant interaction is a 90% CI for the ratio for AUC0-t, AUC0-∞, and Cmax to be within the 0.80 to 1.25 interval, representing a maximum of 20% difference between treatments; Test type: Superiority or Other; ANOVA; Ratio (%) (Test/Reference) = 106.43, 90% CI 2-sided [101.10 to 112.04] — Ratio (theophylline+colchicine/theophylline) of LSMs calculated using the exponentiation of the difference between treatment LSM from the log-transformed AUC(0-∞) , expressed as a percentage relative to the reference treatment

5. Primary Outcome: Apparent Total Body Clearance (CL/F) of Theophylline
Description: Apparent total body clearance after oral administration, calculated as Dose /(AUC0-∞).
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
liters/hour | 1.832 (0.5849) | 1.741 (0.4799)
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Analysis of variance (ANOVA) was performed on the log-transformed CL/F to calculate least squares mean (LSM) for each treatment. The ANOVA model included sequence, treatment, and treatment within a sequence as fixed effects, and participant as a random effect. The criterion for demonstrating a lack of a clinically significant interaction is a 90% CI for the ratio for AUC0-t, AUC0-∞, and Cmax to be within the 0.80 to 1.25 interval, representing a maximum of 20% difference between treatments; Test type: Superiority or Other; ANOVA; Ratio (%) (Test/Reference) = 93.96, 90% CI 2-sided [89.25 to 98.92] — Ratio (theophylline+colchicine/theophylline) of LSMs calculated using the exponentiation of the difference between treatment LSM from the log-transformed CL/F, expressed as a percentage relative to the reference treatment

6. Primary Outcome: Apparent Total Volume of Distribution (Vd/F) of Theophylline
Description: Apparent total volume of distribution after oral administration, calculated as Dose /(AUC0-∞) * Apparent first-order elimination rate constant [Kel])
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Theophylline | Theophylline + Colchicine
Number analyzed (Participants) | 30 | 28
liters | 36.21 (13.03) | 34.44 (10.39)
Statistical Analysis 1: Comparison: Theophylline vs Theophylline + Colchicine; Analysis of variance (ANOVA) was performed on the log-transformed Vd/F to calculate least squares mean (LSM) for each treatment. The ANOVA model included sequence, treatment, and treatment within a sequence as fixed effects, and participant as a random effect. The criterion for demonstrating a lack of a clinically significant interaction is a 90% CI for the ratio for AUC0-t, AUC0-∞, and Cmax to be within the 0.80 to 1.25 interval, representing a maximum of 20% difference between treatments; Test type: Superiority or Other; ANOVA; Ratio (%) (Test/Reference) = 98.59, 90% CI 2-sided [90.97 to 106.85] — Ratio (theophylline+colchicine/theophylline) of LSMs calculated using the exponentiation of the difference between treatment LSM from the log-transformed Vd/F, expressed as a percentage relative to the reference treatment

ADVERSE EVENTS:
Time Frame: From the time of first study drug administration until 5 days after last dose.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Theophylline: Theophylline 300 mg, solution, orally, on Day 1, followed by a 4-day washout period.
- Colchicine: Colchicine, 0.6 mg tablet, orally, twice daily, from Days 5-18.
- Colchicine + Theophylline: Theophylline 300 mg, solution, orally, single dose and colchicine 0.6 mg, tablets, orally, twice daily, on Day 19.
Arm/Group | Theophylline | Colchicine | Colchicine + Theophylline
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 10/30 | 10/30 | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Theophylline (N=30) | Colchicine (N=30) | Colchicine + Theophylline (N=29)
Palpitations (Cardiac disorders) | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Feeling jittery (General disorders) | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 5
Headache (Nervous system disorders) | 2 | 1 | 4
Somnolence (Nervous system disorders) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.